CLINICAL TRIAL: NCT05203224
Title: Improving Early Reperfusion With Adjuvant Dornase Alfa in Large Vessel Ischemic Stroke (EXTEND-IA DNase)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBC2101
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke
Keywords: thrombolysis; thrombolytic; endovascular thrombectomy; tenecteplase; dornase alfa; DNase
MeSH Terms: conditions — Ischemic Stroke | interventions — dornase alfa; Deoxyribonucleases

STUDY DESIGN:
Intervention Model Description: Bayesian Optimised Phase 2 dose-finding umbrella trial
Masking Description: No blinding given single arm study but Independent core laboratory adjudication of the primary outcome, mRS (secondary outcome) performed by central assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenous Dornase alfa (DNase) (Experimental): Patients will receive a single intravenous dose of dornase alfa (at either 0.125mg/kg, 0.25mg/kg, 0.5mg/kg or 1mg/kg in escalating tiers), administered as a bolus over ~30 seconds.
  Interventions: Drug: Dornase Alfa

INTERVENTIONS:
Drug: Dornase Alfa — Intravenous Dornase alfa
  Other Names: DNase; Pulmozyme

SUMMARY:
Patients presenting to the emergency department with acute ischemic stroke, who are are eligible for standard intravenous thrombolytic therapy within 4.5 hours of stroke onset will be assessed for major vessel occlusion to determine their eligibility for the trial. All participants will receive intravenous tenecteplase (or alteplase due to manufacturer shortage) and endovascular thrombectomy as standard care. The trial is a Bayesian Optimised Phase 2 dose-finding umbrella trial (single arm versus objective performance criterion of 20% substantial reperfusion prior to endovascular thrombectomy based on the EXTEND-IA TNK trials NCT02388061, NCT03340493). The aim is to determine the optimal dose of intravenous dornase alfa (recombinant human DNase 1) with sufficient promise to take forward in a seamless phase 2b/3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with acute ischemic stroke eligible, using standard criteria, to receive IV thrombolytics within 4.5 hours of stroke onset
2. Patient's age is ≥18 years
3. Intention to perform endovascular thrombectomy Imaging inclusion criteria
4. Arterial occlusion on CTA or MRA of the ICA, M1, M2 or basilar artery

Exclusion Criteria:

1. Intracranial hemorrhage (ICH) identified by CT or MRI
2. Rapidly improving symptoms at the discretion of the investigator
3. Pre-stroke mRS score of ≥ 4 (indicating previous disability)
4. Hypodensity in >1/3 MCA territory or equivalent proportion of basilar artery territory on non-contrast CT
5. Contraindication to imaging with contrast agents
6. Any terminal illness such that patient would not be expected to survive more than 1 year
7. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
8. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with substantial angiographic reperfusion or absence of retrievable intracranial thrombus at initial angiogram without symptomatic intracerebral hemorrhage | 24 hours post-treatment
  composite outcome of reperfusion on initial angiogram (day 0 - expanded Treatment In Cerebral Infarction [eTICI] 2b-3 or no retrievable intracranial thrombus) and assessment of symptomatic intracerebral hemorrhage on brain imaging 24h post-treatment. eTICI 2b-3 indicates reperfusion of >50% of the initially involved arterial territory.

OTHER OUTCOMES:
modified Rankin Scale (mRS) at 3 months | 3 months post stroke
  ordinal analysis versus EXTEND-IA TNK I & II historical control, adjusted for age and baseline National Institutes of Health Stroke Scale (NIHSS) score. mRS is a functional outcome/disability score from 0 (no disability) to 6 (death). NIHSS is a neurological impairment score from 0 (no deficit) to 42 (death)
modified Rankin Scale (mRS) 0-1 or no change from baseline at 3 months | 3 months post stroke
  versus EXTEND-IA TNK I & II historical control, adjusted for age and baseline NIHSS score
modified Rankin Scale (mRS) 0-2 or no change from baseline at 3 months | 3 months post stroke
  versus EXTEND-IA TNK I & II historical control, adjusted for age and baseline NIHSS score
Proportion of patients with 8 point reduction in NIHSS or reaching 0-1 at 3 days (early neurological improvement) | 3 days post stroke
  versus EXTEND-IA TNK I & II historical control, adjusted for age and baseline NIHSS score
Proportion of patients with near-complete reperfusion (eTICI 2c/3) at conclusion of the endovascular procedure | day 0 (end of endovascular thrombectomy)
  versus EXTEND-IA TNK I & II historical control
Symptomatic intracranial hemorrhage (SICH) | 36 hours post treatment
  Symptomatic intracranial hemorrhage includes any sub-arachnoid bleeding associated with clinical symptoms and symptomatic intracerebral hemorrhage (SICH). SICH is defined as "Intracerebral hemorrhage (parenchymal hematoma type 2 - PH2 within 36 hours of treatment) combined with neurological deterioration leading to an increase of ≥4 points on the NIHSS from baseline, or death"
Death due to any cause | up to 3 months post stroke
  versus EXTEND-IA TNK I & II historical control, adjusted for age and baseline NIHSS

CONTACTS AND LOCATIONS:
Overall Officials: Bruce CV Campbell, MBBS PhD, Principal Investigator — University of Melbourne
Locations (3):
- Australia (3):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient data will be uploaded to the Virtual Stroke Trials Archive (http://www.virtualtrialsarchives.org/vista/) 2 years after the publication of the primary manuscript. Qualified investigators can access data after submission of a project proposal that has been approved by the VISTA steering committee.
Time Frame: 2 years after the publication of the primary manuscript
Access Criteria: Qualified investigators can access data after submission of a project proposal that has been approved by the VISTA steering committee.

REFERENCES:
- [Derived] Di G, Vazquez-Reyes S, Diaz B, Pena-Martinez C, Garcia-Culebras A, Cuartero MI, Moraga A, Pradillo JM, Esposito E, Lo EH, Moro MA, Lizasoain I. Daytime DNase-I Administration Protects Mice From Ischemic Stroke Without Inducing Bleeding or tPA-Induced Hemorrhagic Transformation, Even With Aspirin Pretreatment. Stroke. 2025 Feb;56(2):527-532. doi: 10.1161/STROKEAHA.124.049961. Epub 2025 Jan 27. PMID 39869712